CLINICAL TRIAL: NCT00234936
Title: Quality of Life Study With Adalimumab in Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEXI -P01-03; ESCALAR
Record Dates: First submitted 2005-09-16; First posted 2005-10-10 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2007-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; adalimumab; quality of life
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

INTERVENTIONS:
Drug: Adalimumab
Drug: Methotrexate

SUMMARY:
The purpose of the study is to evaluate the ability of adalimumab combined with methotrexate to improve the quality of life in patients with active RA.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 or older and in good health (Investigator discretion) with a recent stable medical history
* Subject has a diagnosis of rheumatoid arthritis as defined by the 1987 ACR criteria
* Subjects with treatment failure criteria to Mtx or Mtx + another DMARD

Exclusion Criteria:

* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant
* Previous treatment with approved biological agents (etanercept, infliximab, anakinra) in the last 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-12

PRIMARY OUTCOMES:
QOL | 12 months

SECONDARY OUTCOMES:
Patient reported outcomes
Clinical response indicators
Safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott